CLINICAL TRIAL: NCT02238899
Title: Multicenter Register for Children and Young Adults With Intracranial Localized Medulloblastoma, Central Nervous System (CNS)- Primitive Neuroectodermal Tumour (PNET), or Ependymoma
Brief Title: Multicenter Register for Children and Young Adults With Intracranial Localized Medulloblastoma, CNS-PNET or Ependymoma
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: HIT 2000 Interim Register
Record Dates: First submitted 2013-01-18; First posted 2014-09-12 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Medulloblastoma, Childhood; Cerebral Primitive Neuroectodermal Tumor; Ependymoma
MeSH Terms: conditions — Medulloblastoma; Neuroectodermal Tumors, Primitive; Ependymoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tumor material, CSF, and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The Register is based on the study HIT 2000 that recruited patients until 31.12.2011. All german patients with intracranial medulloblastoma, CNS-PNET, ependymoma can be included in the register. Object of the register is to maintain the quality of diagnostic standard by using of central review (Neuroradiology, Pathology, and cranio spinal fluid (CSF) cytology).

Furthermore, the register should enable to continue the collection of epidemiologic data and biological material (tumor material, CSF, and blood) for associated studies.

DETAILED DESCRIPTION:
The Register is based on the study HIT 2000 that recruited patients until 31.12.2011. All german patients with intracranial medulloblastoma, CNS-PNET, ependymoma can be included in the register. Object of the register is to maintain the quality of diagnostic standard by using of central review (Neuroradiology, Pathology, and cranio spinal fluid (CSF) cytology).

Furthermore, the register should enable to continue the collection of epidemiologic data and biological material (tumor material, CSF, and blood) for associated studies.

The register gives recommendations for the therapy of the patients, but these are not mandatory.

ELIGIBILITY:
Inclusion Criteria:

* age at diagnosis 0-21 years
* histologically proven medulloblastoma, CNS-PNET (incl. pineoblastoma, ependymoblastoma, CNS-neuroblastoma), or ependymoma (WHO II/ III)

Exclusion Criteria:

* none

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with medulloblastoma, CNS-PNET (incl. pineoblastoma, ependymoblastoma, CNS-neuroblastoma), or ependymoma (WHO II/ III) and age at diagnosis 0-21 years
Sampling Method: Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Event free survival (EFS) | up to 10 years
  event free survival probability rates will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Rutkowski, Prof., Principal Investigator — University Hospital Hamburg
Locations (1):
- University Hospital, Hamburg, Germany